CLINICAL TRIAL: NCT03858595
Title: Optimizing Gestational Weight Gain, Birth Weight and Other Perinatal Outcomes Among Pregnant Women at Risk of Hypertension in Pregnancy by Regular Monitoring of Weight Gain and Blood Pressure: A Pilot Randomized Controlled Trial
Brief Title: Optimizing Gestational Weight Gain, Birth Weight and Other Perinatal Outcomes Among Pregnant Women at Risk of Hypertension in Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Salu Design Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-18026
Record Dates: First submitted 2018-12-20; First posted 2019-02-28 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-06

CONDITIONS: Hypertension, Pregnancy-Induced; Hypertension, Essential Hypertension; Hypertension; Pre-Eclampsia; Hypertension in Pregnancy
Keywords: Eclampsia,; Pre-Eclampsia; Low birthweight; Wearable; continuous monitoring
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Essential Hypertension; Hypertension; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, two-arm, parallel, and open-label randomized controlled external pilot trial. Eligible participants (high-risk pregnant women) will be individually randomized 1:1 to the intervention arm who will regularly monitor their nutritional status (rate of gestational weight gain) using a digital weighing scale and continuously self-monitor their blood pressure using a wearable device (Salu Health Gauge) from 20 weeks of gestation up to termination of to pregnancy alongside conventional antenatal and postnatal care or the control arm who will receive conventional antenatal and postnatal care only.
Masking Description: Neither the participants nor the investigators or the assessors of outcomes can be blinded to allocation because of the obvious nature and the delivery procedure of the interventions which investigators are going to provide and thus, investigators are obliged to make the RCT non-blinded/open. However, it is prudent to mention that the outcomes of the trial are of objective nature. Furthermore, the randomization, as well as statistical analysis, will be carried out by someone unconnected to the recruitment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Women in the intervention arm will be provided with the "Health Gauge" device. With this device, the women will be able to do self-monitoring of blood pressure as well as a few other things like heart rate, daily activities. Investigators will train our study participants (high-risk pregnant women) on how to use Salu Health Gauge to measure BP as well as how to charge them. Trained FFWs will visit the households weekly and synchronize the device with a tablet computer to collect the stored data. The FFWs will measure the weight of the participants using a digital weighing scale at enrollment and on a monthly bases thereafter. Investigators will keep monitoring up to termination of pregnancy. in any health issue arises, our health worker will ensure that an appropriate referral is made to a tertiary care facility. This intervention will be in addition to the conventional antenatal and postnatal care.
  Interventions: Device: Self monitoring of blood pressure using Health Gauge Device and monthly monitoring of weight gain
- Control group (No Intervention): All those women randomized to the control arm will receive conventional antenatal and postnatal care only. Investigators will collect the outcome data from the households and/or the health centers by follow-up visits or over phone. Investigators will consell participants, women both in the control group, to make at least four antenatal visits. In addition, Investigators will provide counselling about eating healty and keeping physically active during pregnancy. Investigators will provide general nutrition education on taking balanced energy and protein diet.

INTERVENTIONS:
Device: Self monitoring of blood pressure using Health Gauge Device and monthly monitoring of weight gain — Women in the intervention arm will be provided with the "Health Gauge" device. With this device, the women will be able to do self-monitoring of blood pressure as well as a few other things like heart rate, daily activities. We will also measure weight gain of the mothers at monthly basis.
  Arms: Intervention

SUMMARY:
Background:

1. Burden: Hypertensive disorders of pregnancy, including preeclampsia, complicate up to 10% of pregnancies worldwide, constituting one of the greatest causes of fetal growth restriction, preterm birth, low birth weight, perinatal mortality, and maternal morbidity and mortality. In Bangladesh, 24% of all maternal deaths are directly attributed to hypertensive causes. Conventional antenatal care practice often delays in or misses diagnosing hypertension in pregnancy, which makes the women vulnerable to its adverse consequences.
2. Knowledge gap: Although there are randomised controlled trials (RCT) of efforts directed at preventing development of hypertension in pregnancy or reducing its complications, there have been no published RCTs of the intervention focusing on regular monitoring of weight gain and blood pressure among pregnant women who are at risk of developing hypertension in pregnancy or its complications to ensure early diagnosis, and thereby optimizing the perinatal outcomes through prompt referral and management.
3. Relevance: To undertake an RCT of intervention to optimize adverse consequences in hypertension in pregnancy raises important practical concerns including: commitment of the enrolled women, the need to make a decision regarding participation due to longer duration of intervention and adherence to protocol. Investigators aim to perform this study to address whether an RCT of the intervention in individual patients is an appropriate trial design, and is feasible.

Objectives:

1. To evaluate the accuracy of Salu Health Gauge device in measuring blood pressure.
2. To test the design, feasibility, acceptability and fidelity of a future definitive randomized controlled trial focusing on regular monitoring of weight gain and continuous self-monitoring of blood pressure among pregnant women who are at risk of developing hypertension in pregnancy.

Methods:

The study will be completed in two steps: 1) the validation of Salu Health Gauge and 2) the pilot trial. The study will be conducted in Matlab, Bangladesh. Salu Health Gauge device will be validated according to the European Society of Hypertension International Protocol revision 2010 (ESH-IP revision 2010) in general adult population (including men and non-pregnant women) as well as in specific groups such as adolescents and pregnant women. The pilot trial is designed as a prospective, two-arm, parallel, and open-label randomized controlled external pilot trial. Eligible participants (pregnant women at risk of developing hypertension in pregnancy) will be individually randomized 1:1 to the intervention arm who will use a wearable device (Salu Health Gauge) from 20 weeks of gestation up to termination of pregnancy alongside conventional antenatal and postnatal care or the control arm who will receive conventional antenatal and postnatal care only. In Matlab, a woman is diagnosed as pregnant by HDSS field staff by 12-16 weeks of gestation and is enlisted. The investigators will obtain this list from HDSS and conduct baseline interviews to identify pregnant women at risk of developing hypertension in pregnancy.

Outcome measures/variables:

1. Feasibility outcomes: Recruitment rate, Retention rate, compliance, Acceptability etc.
2. Clinical outcomes: gestational weight gain, birth weight, adverse consequence of hypertension in pregnancy (episodes or occurrence and when), blood pressure profile of high-risk pregnancies, prevalence of specific risk factors for hypertension in pregnancy
3. Serious adverse events

DETAILED DESCRIPTION:
Background of the Project including Preliminary Observations Hypertensive disorders of pregnancy, including preeclampsia, complicate up to 10% of pregnancies worldwide, constituting one of the greatest causes of fetal growth restriction, preterm birth, low birth weight, perinatal mortality, and maternal morbidity and mortality.

Odegard et al. found that hypertension in pregnancy, particularly severe and early-onset preeclampsia were associated with significant fetal growth restriction. They showed that preeclampsia was associated with a 5% (95% CI 3%, 6%) reduction in birth weight. In severe preeclampsia, the reduction was 12% (95% CI 9%, 15%), and in early-onset disease, birth weight was 23% (95% CI 18%, 29%) lower than expected. The risk of small-for-gestational-age (SGA) birth was four times higher (relative risk = 4.2; 95% CI 2.2, 8.0) in infants born after preeclampsia.

Pre-eclampsia is also responsible for preterm birth, either spontaneous or through iatrogenic delivery. Lancet Pre-eclampsia series estimated that severe pre-eclampsia increased the risk of preterm delivery by 15-67%, and fetal growth restriction by 10-25%.

Hypertensive disorders of pregnancy are the most common causes of maternal mortality in Europe and are responsible for one-tenth of the maternal deaths in Asia and Africa. Prevalence of preeclampsia, the vilest form of hypertensive disorders of pregnancy, is 12% in Bangladesh. Hypertension in pregnancy or its complications can happen any time during pregnancy, delivery or postnatal period.

Definition and classification of hypertensive disorders in pregnancy Hypertensive disorders of pregnancy are diagnosed by systolic blood pressure (BP) of 140 mmHg or greater and/or diastolic BP of 90 mmHg or greater on at least two occasions more than 4 h apart while resting. Preexisting hypertension may not be evident in the first and second trimesters owing to the physiologic reduction in BP, thus causing confusion with gestational hypertension. Hypertensive disorders of pregnancy or their complications usually manifest after 20 weeks of pregnancy.

The revised International Society for the Study of Hypertension in Pregnancy (ISSHP) classification (2013) for hypertensive disorders in pregnancy is as follows:

1. Chronic hypertension
2. Gestational hypertension
3. Pre-eclampsia - de novo or superimposed on chronic hypertension
4. White coat hypertension

Chronic hypertension Chronic hypertension refers to high blood pressure predating the pregnancy. In practice we rely upon the first trimester blood pressure (measured before 20 weeks of gestation) to define normal or high blood pressure in these women. Most cases of chronic hypertension will be due to essential hypertension, usually accompanied by a family history of hypertension and often by overweight or obesity. Other secondary causes of hypertension are less common and in this age group are usually underlying primary renal parenchymal disorders (such as reflux nephropathy or glomerulonephritis) and less commonly, fibromuscular hyperplasia of the renal arteries or primary hyperaldosteronism.

Gestational hypertension Gestational hypertension is defined as the de novo development of high blood pressure after 20 weeks gestation, without any of the abnormalities that define preeclampsia. This condition is usually benign. However, it can progress to pre-eclampsia in about 25% of cases, more so when the hypertension presents before 32 weeks.

Preeclampsia

The revised ISSHP definition of pre-eclampsia (2014) is:

Hypertension developing after 20 weeks gestation and the coexistence of one or more of the following new onset conditions:

1. Proteinuria
2. Other maternal organ dysfunction:

   * renal insufficiency (creatinine >90 µmol/L)
   * liver involvement (elevated transaminases and/or severe right upper quadrant or epigastric pain)
   * neurological complications (examples include eclampsia, altered mental status, blindness, stroke, or more commonly hyperreflexia when accompanied by clonus, severe headaches when accompanied by hyperreflexia, persistent visual scotomata)
   * haematological complications (thrombocytopenia, DIC, haemolysis)
3. Uteroplacental dysfunction • foetal growth restriction

White-coat hypertension In the general population, up to one in four patients with elevated clinic or office blood pressure have white coat hypertension. This diagnosis can be eliminated partly by having clinic or office blood pressures recorded by a nurse, rather than a doctor, preferably using repeated blood pressure readings. Ideally, the diagnosis is confirmed by demonstrating normal BP using 24 h ambulatory BP monitoring (ABPM) in the first half of pregnancy. There are limited studies on the outcome of these pregnancies but it appears that up to half will develop true gestational hypertension or pre-eclampsia. Increased surveillance is required throughout pregnancy to detect the emergence of pre-eclampsia. Maternal blood pressure should be checked regularly, preferably weekly.

Aetiology and Risk Factors Chronic hypertension occurs in around 20% of women of childbearing age, with the exact prevalence dependent on age, ethnicity, and comorbidities such as diabetes and obesity. The pathophysiologic mechanisms of gestational hypertension are unknown, but are probably the same as those of essential hypertension in the nonpregnant individual, because gestational hypertension increases future post-pregnancy hypertension risk. Gestational hypertension and preeclampsia are separate disease processes with different mechanisms. Evidence supporting this theory includes the differential risk factors, specific histologic changes in the placenta and kidneys associated with preeclampsia only, antiangiogenic peptides of placental origin, the levels of which are elevated in preeclampsia but not in gestational hypertension, and a far lower circulating volume in women with preeclampsia compared with women with gestational hypertension. Table 1 summarizes the risk factors associated with preeclampsia.

Risk factors for preeclampsia

1. Maternal Advanced age (older than 40 years)
2. Black race
3. Interpregnancy interval less than 2 years, or more than 10 years
4. Mother born small for gestational age
5. Nulliparity
6. Preeclampsia or gestational hypertension in a prior pregnancy
7. Chronic hypertension
8. Hyperlipidemia
9. Obesity (BMI ≥35 kg/m2) and insulin resistance
10. Pregestational diabetes mellitus
11. Chronic kidney disease
12. Pre-existing thrombophilia
13. Systemic lupus erythematosus and antiphospholipid syndrome
14. History of migraine
15. Use of SSRIs beyond the first trimester
16. Maternal infections
17. No baseline use of oral contraceptives
18. Polycystic ovarian syndrome
19. Women who have donated a kidney
20. Paternal First pregnancy with partner
21. Limited paternal sperm exposure (<6 months) prior to the pregnancy
22. Partner who fathered a preeclamptic pregnancy in another woman
23. Fetal Multifetal gestation
24. In vitro fertilization
25. Hydropic degeneration of placenta
26. Others Pregnancies after donor insemination, oocyte donation, embryo donation
27. Family history of preeclampsia
28. Family history of coronary heart disease

Pathogenesis of Preeclampsia Although the pathogenesis of pre-eclampsia remains largely unknown, the leading hypotheses strongly rely on disturbed placental function in early pregnancy. However, preeclampsia, including preeclampsia with severe systemic organ involvement and seizures, can first develop in the postpartum period.

Consequences of preeclampsia

Preeclampsia is a major obstetric problem leading to substantial maternal and perinatal morbidity and mortality worldwide, especially in developing countries. Maternal and perinatal outcomes in preeclampsia depend on one or more of the following: gestational age at time of disease onset, severity of disease, quality of management, and presence or absence of pre-existing medical disorders. Maternal and fetal complications in severe preeclampsia are as follows:

Maternal complications

* Abruptio placentae
* Disseminated coagulopathy/HELLP syndrome
* Pulmonary edema/aspiration
* Acute renal failure
* Eclampsia
* Liver failure or hemorrhage
* Stroke
* Death
* Long-term cardiovascular morbidity

Neonatal complications

* Preterm delivery
* Fetal growth restriction
* Hypoxia-neurologic injury
* Stillbirth
* Neonatal death
* Prematurity-associated complications from early delivery
* Long-term cardiovascular morbidity associated with low birthweight

Continuous blood pressure monitoring (CBPM) Hypertension in pregnancy leads to preterm birth, stillbirths, neonatal mortality and maternal death. Therefore, monitoring of blood pressure during and after pregnancy is one of the most important components of antenatal and postnatal care. In conventional antenatal or postnatal care, a single BP measurement at home/clinic is considered to define normal or high blood pressure. But the single measurements at the office/clinics may not reflect the true BP. They may be elevated when the true BP is normal (white coat hypertension) or they may be normal when the true BP is elevated. It becomes more important to have accurate BP measurement when mothers are at risk of gestational hypertension or preeclampsia for early diagnosis to monitor responsiveness to drugs. Therefore, in order to ensure an accurate diagnosis at the earliest, repeated measurement of BP should be taken. One of the ways of taking multiple measurements is 24 hours ambulatory blood pressure monitoring (ABPM).

24 hours of ambulatory blood pressure monitoring (ABPM) 24-hours-Ambulatory blood pressure monitoring (ABPM), which can more precisely characterize changes in BP throughout daily activities, has been found to be superior to clinic BP monitoring in predicting cardiovascular morbidity and mortality. This method nullifies the chance of observer bias and provides a large number of data by performing multiple measurements throughout the day. Ambulatory BP readings may be useful in differentiating primary from secondary hypertension. It is also an important tool to identify white coat hypertension.

ABPM in pregnancy Blood pressure has a property of circadian variation and over the period variation. So in the beginning of pregnancy, BP reduces and in the second trimester (mostly after 20 weeks) it increases again. Elevation of BP is the hallmark for the diagnosis of gestational hypertension and preeclampsia. But conventional practice for measuring BP during the antenatal or postnatal visit at the clinic or home by health workers does not give proper predictive value for hypertensive crisis due to its isolated measurements. Recent studies have found that BP drops during the night in preeclamptic patients.

However, ABPM is not a conventional practice in measurement of BP over a conventional method. BP measurement in pregnancy has relied mostly on a few measurements taken by the physician or health workers. The reason behind this trend is mostly the high cost of ABPM. Additionally, it is not available in all the places in the world. Even after getting this at a high price, ABPM cannot be used for several days due to weight and discomfort in using it day and night. Finally, there are no unanimous guidelines that suggest a particular time of using it during pregnancy. Some of the studies used it in the first trimester and a few tried in the second trimester. One of them investigated after every 4 weeks to monitor the BP in the aim of predicting the hypertensive crisis in compare to traditional BP measurements.

Continuous blood pressure monitoring (CBPM) with wrist devices Efforts have been made to establish accurate methods for continuously monitoring blood pressure based on other physiological parameters. Blood pressure is often estimated by means of linear models, in which the variables are the extracted parameters from ECG and PPG, representing the response of the cardiovascular system. Among them mostly used parameters are Pulse transmit time (PTT) along with pulse amplitude, heart rate and pulse width (PW). PW is more sensitive to changes in systemic vascular resistance (SVR) than other indices of pulse wave. The SVR is determined by changes in artery diameter or changes in blood viscosity. Changes in PW provide valuable evidence with respect to changes in pulse wave velocity (PWV) too.

Several models have been developed to estimate SBP and DBP, and studies have identified PW as a better estimator than PTT. Additionally, to estimate BP using PW does not require ECG recording which is mandatory for PTT. The correlation is also higher between measured and estimated BP using PW.

Justification of the study In 2012, an estimated 23.3 million infants were born small for gestational age in low and middle-income countries. The incidence of fetal growth restriction in Bangladesh, manifested by SGA births, is among the highest in the world. The prevalence of SGA in Bangladesh has been estimated to be about 30.5%. The rate of preterm birth is high as well, which is at 14.1%. Reducing the burden of SGA births and malnutrition in children under five years in Bangladesh and other LMICs is now one of the major concerns of the governments and many international agencies. However, the most tractable pathways for effective interventions to promote healthy fetal growth remain unclear.

According to the Bangladesh Maternal Mortality Survey (BMMS) 2010, maternal mortality declined from 322 in 2001 to 194 in 2010, a decline of about 40 percent. The average rate of decline was about 3.3 percent per year. Although Bangladesh did a laudable job in reducing maternal mortality up until 2010, the MMR has stalled thereafter. The MMR estimate from the BMMS 2016 is 196 maternal deaths per 100,000 live births, almost identical to the estimate of BMMS 2010.

Hypertensive disorders in pregnancy and their complications are the second most important causes of maternal death. In conventional practice, pregnant women are checked for high BP or its complications during antenatal visits. Antenatal care (ANC) visit rate has increased considerably in Bangladesh. In 2014, 78% of the expectant mothers received at least one ANC visit and about 31% received 4 or more whereas, in 2000, it was 34% and 10.5% respectively. However, this improvement in maternal health-seeking behavior has not translated into a further reduction of maternal deaths. Increasing facility delivery is important but not sufficient to lower MMR. Quality of care is fundamental to improve maternal health outcomes. Several studies in other countries have highlighted the importance of the quality of care in translating the use of maternal health services into improved health outcomes. The quality of health care is generally poor in Bangladesh.

The cause-specific mortality ratio due to eclampsia increased from 39 per 100,000 live births in 2010 to 46 per 100,000 live births in 2016. There has been little progress in interventions to address this issue.

As blood pressure has a property of circadian variation and over the period variation, and current practice of measuring blood pressure, which is subject to interpersonal and digit/number bias, results in misdiagnosis of hypertension in pregnancy.

A better way of diagnosing hypertension in women can be by taking multiple measurements through continues monitoring of blood pressure. ABPM could be an option, but it is also subject to discomfort and limitation of only 24 to 48 hours of continuous monitoring. A novel way of continuous monitoring of blood pressure is by using ECG and PPG measuring both PW and PTT. Salu Health Gauge is a device that uses PW and PPT to measure blood pressure and can store and give a picture of blood pressure variability over the time for a very long period.

Other methods such as uterine artery Doppler artery ultrasonography, maternal blood concentrations of angiogenic factors and metabolomics are also available to predict and monitor hypertension in pregnancy. However, these tools are further expensive and inconvenient for resource-poor settings like Bangladesh. A self-used wearable device would be a better choice for monitoring among women at risk of hypertension in pregnancy.

Although there are randomized controlled trials (RCT) of efforts directed at preventing development of hypertension in pregnancy or reducing its complications, there have been no published RCTs of the intervention focusing on regular monitoring of weight gain and blood pressure among pregnant women who are at risk of developing hypertension in pregnancy or its complications to ensure early diagnosis, and thereby optimizing the gestational weight gain, birth weight and other perinatal outcomes through prompt referral and management.

To undertake an RCT of an intervention to optimize adverse consequences in hypertension in pregnancy raises important practical concerns including commitment of the enrolled women, the need to make a decision regarding participation due to longer duration of intervention and adherence to protocol. The investigators aim to perform this study to address whether an RCT of the intervention in individual patients is an appropriate trial design, and is feasible with regard to i) maternal recruitment and retention ii) participant acceptability, iii) adherence to protocol. In addition, investigators wish to estimate the incidence of hypertension in pregnancy and its adverse consequences in the study population.

Specific Objective of the Validation Studies:

1. To evaluate the accuracy of Salu Health Gauge device (wrist-worn) in measuring blood pressure (BP), which is useful for continuous self-monitoring of BP, in general adult population (including men and non-pregnant women) as well as in specific groups such as adolescents and pregnant women, according to the European Society of Hypertension International Protocol revision 2010 (ESH-IP revision 2010)

Specific Objectives of the Pilot Trial:

The aims of this pilot trial are to test the design and methods of a future definitive randomized controlled trial and examine the feasibility, acceptability and fidelity of the intervention focusing on regular monitoring of rate of gestational weight gain using a digital weighing scale and continuous self-monitoring of blood pressure using a wearable device (Salu Health Gauge) among pregnant women who are at risk of developing hypertension in pregnancy or its complications to ensure early diagnosis, and thereby optimizing the gestational weight gain, birth weight and other perinatal outcomes through prompt referral and management. The specific objectives of this pilot trial are:

1. To obtain reliable estimates of eligibility, consenting, response and attrition rates and level of missing data
2. To determine whether the eligibility criteria are too open or too restrictive by assessing the proportion of participants actually developing outcomes, and to explore the variability of the risk factors
3. To assess the appropriateness (and factors inﬂuencing this) of the clinical outcome measures as methods to measure the efficacy of the intervention within a definitive trial, and to explore the variability of the clinical outcomes in terms of type and time of occurring
4. To investigate the acceptability of the intervention in terms of compliance and adherence to the intervention schedule, and the contextual factors associated with variation
5. To assess the feasibility and acceptability of recruitment, randomization, allocation concealment and outcome assessment procedures
6. To evaluate the feasibility of regular monitoring of the rate of gestational weight gain using a digital weighing scale to optimize gestational weight gain, birth weight and other perinatal outcomes
7. To evaluate the functionality and usability of the Salu Health Gauge device with a particular focus on the feasibility of storage, collection, and analysis of complete blood pressure profile
8. To evaluate participant satisfaction with using the device during the prenatal period
9. To conduct a process evaluation to assess the intervention fidelity in terms of adherence to the intervention manual by participants and trainers
10. To evaluate resource use and costs associated with intervention delivery and outcome measurement, and to assess the feasibility of using existing health facility and other resources
11. To explore the occurrence of any adverse event or unintended consequences of the intervention
12. To collect and synthesize data, from which the sample size of a definitive trial could be estimated
13. To measure the variances and point and interval estimates for the clinical outcomes, and 95% confidence intervals for the diﬀerence between the arms
14. To evaluate the appropriateness of the trial procedures, design, and duration, and to explore the potential effect of the intervention to determine whether this suggests a clinically important effect which will support the conduct of a definitive trial

Research Design and Methods

The study will be completed in two steps, which are described in detail as follows:

Step 1: The Validation Studies

The "Health Gauge" device investigators will use in our study is made by Salu Design located in Alberta, Canada. Salu Design has found that, in internal quality control, the "Health Gauge" device gives precise and accurate blood pressure (BP) measurement in adults (personal communication, Randy Duguay, Salu design, Alberta, Canada). However, it is important to ensure that the device is functioning accurately in our setting. This validation study aims to evaluate the accuracy of the device according to the European Society of Hypertension International Protocol revision 2010 (ESH-IP revision 2010). The investigators will do the validation of the "Health Gauge" device separately for general adult population (including men and non-pregnant women), and for specific groups such as adolescents and pregnant women. The methods and procedures for the validation studies, according to the ESH-IP revision 2010, are described below in brief Salu Health Gauge (wrist-worn) The Salu Health Gauge solution (wrist-worn) provides the world's first compact wrist-based, cuffless heart health management system using a unique combination of 2-contact Electrocardiography (ECG), and Photoplethysmography (PPG), a combination of pulse wave analysis algorithms, machine learning, and neural network computing techniques. The Health Gauge device can simultaneously capture a digitized pulsewave and electrocardiogram signal focusing on the radial artery. When the user touches the outer conductive pad, the solution captures full pulse and ECG signals within seconds, which then provides for calculated blood pressure results, pulse-wave velocity (PWV), and spO2 levels which will be recorded at that moment within 20 seconds. It creates a triangle by connecting two parts of the body (here two hands) and passed through the heart to assess the electric impulses exerted from the heart. The device keeps those measure records in its memory. These data can be synchronized with and accessed from a tablet computer.

Sample size and selection of participants In accordance with the ESH-IP revision 2010, a total of 33 participants who fulfill the age, sex, entry BP and other requirements will be included in the validation study (for general adult population), such as: age ≥25 years, with at least 10 men and 10 women, and 10-12 participants in each of the three BP recruitment ranges: 90-129, 130-160, and 161-180 mmHg for systolic BP (SBP) and 40-79, 80-100, and 101-130 mmHg for diastolic BP (DBP). According to the ESH-IP revision 2010, validation studies in specific groups such as pregnant women will be carried out with necessary modification of these requirements, and all such changes or additions will be clearly described during reporting. All the participants will be recruited from outpatients of Matlab hospital of icddr,b or as volunteers residing in Matlab near Matlab hospital. For validation among the adolescents and pregnant population, the same protocol with slight necessary modifications will be used.

Procedures For BP measurement, the validation team will consist of three persons (two observers and a supervisor) having experience in BP measurements and will be trained by the British and Irish Hypertension Society (BIHS)'s online program.

The gold standard instruments for BP measurement will consist of two standard mercury sphygmomanometers and a good quality double stethoscope. Simultaneous auscultations will be performed by two observers using the double stethoscope (Y tube) and then the BP will be measured. These two observers will be blinded to each other's readings, and the third observer will serve as a supervisor and check the BP readings of the other two observers. The supervisor will make sure that the difference between the two observers is no more than 4 mmHg for SBP and DBP values. Otherwise, the measurement will be repeated.

The participants will be seated in a quiet room with a comfortable room temperature. They will be instructed to avoid talking during the procedure. BP measurements will start after 15 min of rest. The participants will sit with their legs uncrossed and feet flat on the floor in a chair with a supportive back, as well as elbow and forearm rest.

The BP measurements will be alternated between the mercury sphygmomanometer and the Salu Health Gauge device. In total, nine consecutive BP measurements will be performed in each subject using the mercury sphygmomanometers (five times) and the tested device (four times), and will be recorded as follows:

1. Entry BPA with a mercury sphygmomanometer by observers 1 and 2 (used to separate the patients into appropriate BP range groups)
2. BPB by supervisor (device detection BP)
3. BP1 by observers 1 and 2 with a mercury sphygmomanometer
4. BP2 by the supervisor with the test device
5. BP3 by observers 1 and 2 with a mercury sphygmomanometer
6. BP4 by the supervisor with the test device
7. BP5 by observers 1 and 2 with a mercury sphygmomanometer
8. BP6 by the supervisor with the test device
9. BP7 by observers 1 and 2 with a mercury sphygmomanometer

Statistical analysis plan Results will be analyzed and expressed according to the ESH-IP revision 2010 requirements to conclude if the device passes or fails to pass the validation protocol. Details of the analysis procedure have been described elsewhere. In brief, the differences between the test devices and the control measurements will be classified according to whether their values are within 5, 10, or 15 mmHg. The differences will be calculated by subtracting the observer measurement from the test device measurement and classified separately for SBP and DBP. The mean of each pair of observer measurements will be calculated, which is denoted as observer measurement BP1, BP3, BP5, or BP7. Each device measurement will be flanked by two of these observer measurements, and one of them will be selected as the comparative measurement. From these, further measurements will be derived as follows: (a) the differences between BP2 and BP1, BP2, and BP3, BP4 and BP3, BP4 and BP5, BP6 and BP5, and BP6 and BP7 will be calculated; (b) the absolute values of the differences will be calculated; (c) values will be paired according to the device reading; (d) if the values in a pair are unequal, the observer measurement corresponding to the smaller difference will be used; and (e) if the values in a pair are equal, the first of the two observer measurements will be used.

Step 2: The Pilot Randomized Controlled Trial

The pilot trial will commence after the Salu Health Gauge will have passed the validation stage. The "CONSORT 2010 statement: extension to randomized pilot and feasibility trials" recommendations have been followed in preparing this protocol for the pilot randomized controlled trial.

Study design This study is designed as a prospective, two-arm, parallel, and open-label randomized controlled external pilot trial. Eligible participants (high-risk pregnant women) will be individually randomized 1:1 to the intervention arm who will regularly monitor their nutritional status (rate of gestational weight gain) using a digital weighing scale and continuously self-monitor their blood pressure using a wearable device (Salu Health Gauge) from 20 weeks of gestation up to termination of to pregnancy alongside conventional antenatal and postnatal care or the control arm who will receive conventional antenatal and postnatal care only.

Study site The study will be conducted in rural Bangladesh at Matlab, a low-lying riverine area, situated 55 km southeast of the capital of Bangladesh. Since 1966, icddr,b has been running an internationally recognized and unique Health and Demographic Surveillance System (HDSS) involving all 142 villages of the Matlab Upazila, comprising a population of 230,000 people. Registration of vital events like births, deaths, marriages, migration is updated by community health research workers on a bi-monthly basis. Information on reproductive health outcome, contraceptive use, breastfeeding, and immunization have also been collected.

Screening and identification of potentially eligible participants In Matlab, a woman is diagnosed as pregnant by HDSS field staff by 12-16 weeks of gestation and is enlisted. The investigators will obtain this list from HDSS and conduct baseline interviews to identify the high-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* High risk pregnancy
* At 12-16 weeks of gestation
* Aged between 15 to 50 years
* Living in Matlab bangladesh

Exclusion Criteria:

* Have congenital malformation/anomaly in current pregnancy
* Current pregnancy have chromosomal abnormality e.g. Down syndrome
* Have chronic debilitating illness
* Mother is a known case of psychosis
* Who do not have electricity at their house
* Do not have smart phone at their house

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Our study aimed to prevent hypertensive disorders of pregnancy. So only female can be enrolled in the study as participant due to their ability to be pregnant
Enrollment: 70 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Recruitment rate is defined as number of participants recruited per month on average. This outcome is important because unforeseen enrolment challenges are crucial to identify in a pilot RCT.
Retention rate | Till the follow-up period (from 20 weeks to until delivery or termination of the pregnancy) ends
  Retention rate is defined as the proportion of participants who will fully participate in the study until follow-up period (from 20 week up to the delivery) ends.
Adherence to protocol (compliance) | 5 months
  Adherence is defined as the proportion of participants following the intervention protocol. There may be a number of reasons why the participant do not follow the intervention protocol properly. FFWs will enquire the reasons during weekly visits and note the causes and the number of times they have violated the protocol in a log sheet. Understandable protocol deviations (e.g., participant died) will be distinguished from protocol violations (e.g., participant removed the wearable gauge).
Acceptability of the device | 5 months
  Participant acceptability of the device as intervention will be assessed two times during the follow-up period using a Likert scale with 5 level of qualitative response as well as by asking qualitative questions. The quantitative result will be reported as median (interquartile range) score for combined and period specific outcomes. They will be assessed once during the third trimester and in the end of the study. The qualitative part will be reported narratively. up period using a Likert scale as well as by asking qualitative questions. The quantitative result will be reported as median (interquartile range) score for combined and period specific outcome. They will be assessed once during the second trimester, once during the third trimester and finally once during the postnatal period. The qualitative part will be reported narratively.
Acceptability of the BP measurement | 5 months
  Participant acceptability of the BP measurement procure as a part of the intervention will be assessed two times during the follow-up period using a Likert scale with 5 level of qualitative response as well as by asking qualitative questions. The quantitative result will be reported as median (interquartile range) score for combined and period specific outcomes. They will be assessed once during the third trimester and in the end of the study. The qualitative part will be reported narratively.

SECONDARY OUTCOMES:
Rate of gestational weight gain | 20 week of gestation up to termination of pregnancy
  The investigators will measure the gestational weight gain by using increase of maternal weight per month and increase of maternal weight per week. Weight will be measured in kilograms.
Birth weight | 20 week of gestation up to termination of pregnancy
  The investigators will record birth weight in every viable births and will record in grams (gm). Then investigators will compare the birth weight between two groups.
Adverse consequence of hypertension in pregnancy | 20 week of gestation up to termination of pregnancy
  The investigators will measure the adverse consequences of pregnancy due to hypertension during pregnancy. The investigators will record all the episodes or occurrence of adverse events. This will compared in descriptive nature and compare between groups. Adverse events will be for mothers are: abruptio placenta, Disseminated coagulopathy, Pulmonary oedema/aspiration, acute renal failure, eclampsia, liver failure or hemorrhage, stroke, death. Fetal events like intrauterine death/stillbirth, preterm birth, small-for-gestational age, low birth weight, Hypoxia-neurologic injury, neonatal death, complications associated with LBW or preterm births
Blood pressure profile of high risk pregnancies | 20 week of gestation up to termination of pregnancy
  The investigators will motivate mothers to measure blood pressure in mm/Hg for at least six times in a day. Then investigators will prepare a complete profile of blood pressure for her pregnancy from 20 weeks of gestation up to the termination of pregnancy for each participants in intervention groups. The investigators will also make a profile of blood pressure among control groups with their recorded data measured by their respective health professionals (doctors and health workers). The investigators will take the average and compare the blood pressure in different time periods.
Heart rate profile of high risk pregnancies | 20 week of gestation up to termination of pregnancy
  The investigators will motivate the mothers to measure the heart rate for 6 times a day with the health Gauge device. Then heart rate will be calculated in beats per minutes.
Rate of daily activity | 20 week of gestation up to termination of pregnancy
  The investigators will measure the daily activity of pregnant mothers who are at risk of hypertension by step counts per day during their observation period.
Sleeping status of mothers | 20 week of gestation up to termination of pregnancy
  The investigators will take data related to sleeping status of mothers and will be recorded as number of hours passed in different stages of sleeps. The investigators will make a profile for those mothers have higher risk for pregnancy related hypertension
Sociodemographic profile | 6 months
  The investigators will take the data of those mothers enrolled in the study related to their sociodemographic status.

CONTACTS AND LOCATIONS:
Locations (1):
- Icddr,B, Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen S, Irgens LM, Albrechtsen S, Dalaker K. Predicting preeclampsia in the second pregnancy from low birth weight in the first pregnancy. Obstet Gynecol. 2000 Nov;96(5 Pt 1):696-700. doi: 10.1016/s0029-7844(00)01008-5. PMID 11042303
- [Background] Odegard RA, Vatten LJ, Nilsen ST, Salvesen KA, Austgulen R. Preeclampsia and fetal growth. Obstet Gynecol. 2000 Dec;96(6):950-5. PMID 11084184
- [Background] Mol BWJ, Roberts CT, Thangaratinam S, Magee LA, de Groot CJM, Hofmeyr GJ. Pre-eclampsia. Lancet. 2016 Mar 5;387(10022):999-1011. doi: 10.1016/S0140-6736(15)00070-7. Epub 2015 Sep 2. PMID 26342729
- [Background] Sibai B, Dekker G, Kupferminc M. Pre-eclampsia. Lancet. 2005 Feb 26-Mar 4;365(9461):785-99. doi: 10.1016/S0140-6736(05)17987-2. PMID 15733721
- [Background] Kintiraki E, Papakatsika S, Kotronis G, Goulis DG, Kotsis V. Pregnancy-Induced hypertension. Hormones (Athens). 2015 Apr-Jun;14(2):211-23. doi: 10.14310/horm.2002.1582. PMID 26158653
- [Background] Tranquilli AL, Dekker G, Magee L, Roberts J, Sibai BM, Steyn W, Zeeman GG, Brown MA. The classification, diagnosis and management of the hypertensive disorders of pregnancy: A revised statement from the ISSHP. Pregnancy Hypertens. 2014 Apr;4(2):97-104. doi: 10.1016/j.preghy.2014.02.001. Epub 2014 Feb 15. No abstract available. PMID 26104417
- [Background] Jahan M, Hasanuzzaman M, Mahbuba S, Jahan H, Chowdhury S, Ahsan GU, et al. [225-POS]: Prevalence of preeclampsia in pre-gestational diabetic pregnancy in Bangladeshi patients. Pregnancy Hypertension: An International Journal of Women's Cardiovascular Health. 2015;5(1):113-4.
- [Background] Preeclampsia Foundation [cited 2018 1st April]. Available from: https://www.preeclampsia.org/health-information/faqs
- [Background] Vest AR, Cho LS. Hypertension in pregnancy. Curr Atheroscler Rep. 2014 Mar;16(3):395. doi: 10.1007/s11883-013-0395-8. PMID 24477794
- [Background] Zhang J, Zeisler J, Hatch MC, Berkowitz G. Epidemiology of pregnancy-induced hypertension. Epidemiol Rev. 1997;19(2):218-32. doi: 10.1093/oxfordjournals.epirev.a017954. PMID 9494784
- [Background] Saudan P, Brown MA, Buddle ML, Jones M. Does gestational hypertension become pre-eclampsia? Br J Obstet Gynaecol. 1998 Nov;105(11):1177-84. doi: 10.1111/j.1471-0528.1998.tb09971.x. PMID 9853766
- [Background] Franklin SS, Thijs L, Hansen TW, O'Brien E, Staessen JA. White-coat hypertension: new insights from recent studies. Hypertension. 2013 Dec;62(6):982-7. doi: 10.1161/HYPERTENSIONAHA.113.01275. Epub 2013 Sep 16. No abstract available. PMID 24041952
- [Background] Brown MA, Buddle ML, Martin A. Is resistant hypertension really resistant? Am J Hypertens. 2001 Dec;14(12):1263-9. doi: 10.1016/s0895-7061(01)02193-8. PMID 11775136
- [Background] Brown MA, Mangos G, Davis G, Homer C. The natural history of white coat hypertension during pregnancy. BJOG. 2005 May;112(5):601-6. doi: 10.1111/j.1471-0528.2004.00516.x. PMID 15842284
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363
- [Background] Ferrer RL, Sibai BM, Mulrow CD, Chiquette E, Stevens KR, Cornell J. Management of mild chronic hypertension during pregnancy: a review. Obstet Gynecol. 2000 Nov;96(5 Pt 2):849-60. doi: 10.1016/s0029-7844(00)00938-8. PMID 11094241
- [Background] Baguet JP. Out-of-office blood pressure: from measurement to control. Integr Blood Press Control. 2012;5:27-34. doi: 10.2147/IBPC.S30409. Epub 2012 May 16. PMID 22654523
- [Background] Grossman E. Ambulatory blood pressure monitoring in the diagnosis and management of hypertension. Diabetes Care. 2013 Aug;36 Suppl 2(Suppl 2):S307-11. doi: 10.2337/dcS13-2039. No abstract available. PMID 23882064
- [Background] James PR, Nelson-Piercy C. Management of hypertension before, during, and after pregnancy. Heart. 2004 Dec;90(12):1499-504. doi: 10.1136/hrt.2004.035444. No abstract available. PMID 15547046
- [Background] Metoki H, Ohkubo T, Kikuya M, Asayama K, Obara T, Hara A, Hirose T, Hashimoto J, Totsune K, Hoshi H, Satoh H, Imai Y. Prognostic significance of night-time, early morning, and daytime blood pressures on the risk of cerebrovascular and cardiovascular mortality: the Ohasama Study. J Hypertens. 2006 Sep;24(9):1841-8. doi: 10.1097/01.hjh.0000242409.65783.fb. PMID 16915034
- [Background] Flynn JT. Differentiation between primary and secondary hypertension in children using ambulatory blood pressure monitoring. Pediatrics. 2002 Jul;110(1 Pt 1):89-93. doi: 10.1542/peds.110.1.89. PMID 12093951
- [Background] Sheppard JP, Holder R, Nichols L, Bray E, Hobbs FD, Mant J, Little P, Williams B, Greenfield S, McManus RJ. Predicting out-of-office blood pressure level using repeated measurements in the clinic: an observational cohort study. J Hypertens. 2014 Nov;32(11):2171-8; discussion 2178. doi: 10.1097/HJH.0000000000000319. PMID 25144295
- [Background] Haney A, Buysse DJ, Okun M. Sleep and pregnancy-induced hypertension: a possible target for intervention? J Clin Sleep Med. 2013 Dec 15;9(12):1349-56. doi: 10.5664/jcsm.3290. PMID 24340300
- [Background] Staessen JA, Thijs L, Fagard R, O'Brien ET, Clement D, de Leeuw PW, Mancia G, Nachev C, Palatini P, Parati G, Tuomilehto J, Webster J. Predicting cardiovascular risk using conventional vs ambulatory blood pressure in older patients with systolic hypertension. Systolic Hypertension in Europe Trial Investigators. JAMA. 1999 Aug 11;282(6):539-46. doi: 10.1001/jama.282.6.539. PMID 10450715
- [Background] Cohen DL, Townsend RR. Should all patients have ambulatory blood pressure monitoring performed to validate the diagnosis of hypertension? J Clin Hypertens (Greenwich). 2015 May;17(5):412-3. doi: 10.1111/jch.12527. Epub 2015 Mar 10. No abstract available. PMID 25758101
- [Background] Ayala DE, Hermida RC. Ambulatory blood pressure monitoring for the early identification of hypertension in pregnancy. Chronobiol Int. 2013 Mar;30(1-2):233-59. doi: 10.3109/07420528.2012.714687. Epub 2012 Sep 24. PMID 23006127
- [Background] Arza A, Lázaro J, Gil E, Laguna P, Aguiló J, Bailon R, editors. Pulse transit time and pulse width as potential measure for estimating beat-to-beat systolic and diastolic blood pressure. Computing in Cardiology Conference (CinC), 2013; 2013: IEEE.
- [Background] Wu C-M, Chuang CY, Chen Y-J, Chen S-C. A new estimate technology of non-invasive continuous blood pressure measurement based on electrocardiograph. Advances in Mechanical Engineering. 2016;8(6):1687814016653689.
- [Background] Gesche H, Grosskurth D, Kuchler G, Patzak A. Continuous blood pressure measurement by using the pulse transit time: comparison to a cuff-based method. Eur J Appl Physiol. 2012 Jan;112(1):309-15. doi: 10.1007/s00421-011-1983-3. Epub 2011 May 10. PMID 21556814
- [Background] Lee AC, Kozuki N, Cousens S, Stevens GA, Blencowe H, Silveira MF, Sania A, Rosen HE, Schmiegelow C, Adair LS, Baqui AH, Barros FC, Bhutta ZA, Caulfield LE, Christian P, Clarke SE, Fawzi W, Gonzalez R, Humphrey J, Huybregts L, Kariuki S, Kolsteren P, Lusingu J, Manandhar D, Mongkolchati A, Mullany LC, Ndyomugyenyi R, Nien JK, Roberfroid D, Saville N, Terlouw DJ, Tielsch JM, Victora CG, Velaphi SC, Watson-Jones D, Willey BA, Ezzati M, Lawn JE, Black RE, Katz J; CHERG Small-for-Gestational-Age-Preterm Birth Working Group. Estimates of burden and consequences of infants born small for gestational age in low and middle income countries with INTERGROWTH-21st standard: analysis of CHERG datasets. BMJ. 2017 Aug 17;358:j3677. doi: 10.1136/bmj.j3677. PMID 28819030
- [Background] Ashworth A. Effects of intrauterine growth retardation on mortality and morbidity in infants and young children. Eur J Clin Nutr. 1998 Jan;52 Suppl 1:S34-41; discussion S41-2. PMID 9511018
- [Background] Mata LJ, Kromal RA, Urrutia JJ, Garcia B. Effect of infection on food intake and the nutritional state: perspectives as viewed from the village. Am J Clin Nutr. 1977 Aug;30(8):1215-27. doi: 10.1093/ajcn/30.8.1215. PMID 888779
- [Background] General Economics Division (GED). Bangladesh Planning Commission. (2015). Millennium Development Goals: Bangladesh Progress Report 2015. Available from: http://www.plancomm.gov.bd/wp-content/uploads/2015/09/MDGs-Bangladeh-Progress-Report_-PDF_Final_September-2015.pdf. 2015
- [Background] NIPORT. Bangladesh Maternal Mortality and Health Care Survey 2016. 2016;Preliminary report.
- [Background] Brown MA. Is there a role for ambulatory blood pressure monitoring in pregnancy? Clin Exp Pharmacol Physiol. 2014 Jan;41(1):16-21. doi: 10.1111/1440-1681.12106. PMID 23651133
- [Background] O'Brien E, Atkins N, Stergiou G, Karpettas N, Parati G, Asmar R, Imai Y, Wang J, Mengden T, Shennan A; Working Group on Blood Pressure Monitoring of the European Society of Hypertension. European Society of Hypertension International Protocol revision 2010 for the validation of blood pressure measuring devices in adults. Blood Press Monit. 2010 Feb;15(1):23-38. doi: 10.1097/MBP.0b013e3283360e98. No abstract available. PMID 20110786
- [Background] How to measure Blood Pressure. BP Measurement. British and Irish Hypertension Society. https://bihsoc.org/resources/bp-measurement/measure-blood-pressure/. 2017.
- [Background] O'Brien E, Pickering T, Asmar R, Myers M, Parati G, Staessen J, Mengden T, Imai Y, Waeber B, Palatini P, Gerin W; Working Group on Blood Pressure Monitoring of the European Society of Hypertension. Working Group on Blood Pressure Monitoring of the European Society of Hypertension International Protocol for validation of blood pressure measuring devices in adults. Blood Press Monit. 2002 Feb;7(1):3-17. doi: 10.1097/00126097-200202000-00002. No abstract available. PMID 12040236
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394
- [Derived] Hasan SMT, Ahmed SI, Khan MA, Sarker SA, Ahmed T. Achieving Optimal Gestational Weight Gain, Birth Weight, and Perinatal Outcomes Among Pregnant Women at Risk of Hypertension: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 15;9(6):e16676. doi: 10.2196/16676. PMID 32459639